CLINICAL TRIAL: NCT05975099
Title: A Phase 1/2, Randomized, Observer-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Safety and Immunogenicity of Heptavalent mRNA-1975 (SR1-7) and Monovalent mRNA-1982 (SR1) in Parallel Against Lyme Disease in Healthy Participants 18 Through 70 Years of Age
Brief Title: A Study to Evaluate the Safety and Immunogenicity of mRNA-1975 and mRNA-1982 Against Lyme Disease in Participants 18 Through 70 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mRNA-1975/1982-P101
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lyme Disease
Keywords: mRNA-1975; mRNA-1982; Vaccine; Lyme Disease Vaccine; Messenger RNA; Moderna
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- mRNA-1975: Dose 1 (Experimental): Participants will receive 3 intramuscular (IM) injections of the mRNA-1975 vaccine at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1975
- mRNA-1975: Dose 2 (Experimental): Participants will receive 3 IM injections of the mRNA-1975 vaccine at Dose level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1975
- mRNA-1975: Dose 3 (Experimental): Participants will receive 3 IM injections of the mRNA-1975 vaccine at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1975
- mRNA-1975: Dose 4 (Experimental): Participants will receive 3 IM injections of the mRNA-1975 vaccine at Dose level 4 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1975
- mRNA-1982: Dose 1 (Experimental): Participants will receive 3 IM injections of the mRNA-1982 vaccine at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1982
- mRNA-1982: Dose 2 (Experimental): Participants will receive 3 IM injections of the mRNA-1982 vaccine at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1982
- mRNA-1982: Dose 3 (Experimental): Participants will receive 3 IM injections of the mRNA-1982 vaccine at Dose level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1982
- Placebo (Placebo Comparator): Participants will receive 3 IM injections of vaccine-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1975 — Dispersion delivered IM
  Other Names: SR1-7
  Arms: mRNA-1975: Dose 1; mRNA-1975: Dose 2; mRNA-1975: Dose 3; mRNA-1975: Dose 4
Biological: mRNA-1982 — Dispersion delivered IM
  Other Names: SR1
  Arms: mRNA-1982: Dose 1; mRNA-1982: Dose 2; mRNA-1982: Dose 3
Biological: Placebo — Solution delivered IM
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity in parallel of heptavalent mRNA-1975 and monovalent mRNA-1982 against Lyme disease in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 to 39 kilograms/square meter (inclusive) at the Screening Visit.
* Participants of nonchildbearing potential may be enrolled in the study.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy during the study intervention period, and agreement to continue adequate contraception or abstinence through 3 months following last study injection.

Exclusion Criteria:

* Have chronic illness related to Lyme disease or an active symptomatic Lyme disease infection as suspected or diagnosed by a physician.
* Received treatment for Lyme disease within the prior 3 months.
* Had previous vaccination against Lyme disease or participated in the past in any vaccine study for Lyme disease.
* Had a tick bite within 4 weeks prior to the study injection visit.
* Dermatologic conditions that could affect local solicited AR assessments (for example, tattoos; psoriasis patches affecting skin over the deltoid areas).
* Received systemic immunosuppressants for >14 days in total within 180 days prior to the Screening Visit (for corticosteroids, ≥10 milligrams/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study.
* History of myocarditis, pericarditis, or myopericarditis regardless of the timing of past medical history.
* History of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine or intervention that includes one or more of the same components contained in the study injection.
* Has received systemic immunoglobulins, long-acting biological therapies that affect immune responses (for example, infliximab) or blood products within 90 days prior to the Screening Visit or plans to receive them during the study.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 175 (7 days after each study injection)
Number of Participants With Unsolicited Adverse Events (AEs) | Up to Day 196 (28 days after each study injection)
Number of Participants With Medically Attended AEs | Day 1 through Day 337 (6 months after the last study injection)
Number of Participants with AEs of Special Interest, Serious AEs, and AEs Leading to Discontinuation of Study Injection or Study Participation | Day 1 through Day 505 (End of Study)

SECONDARY OUTCOMES:
Geometric Mean Concentration of Anti-outer Surface Protein A (anti-OspA) Binding Immunoglobulin G (IgG) Antibodies Measured by Enzyme-linked Immunosorbent Assay or a Similar Method | Days 1, 29, 85, and 197
Geometric Mean Fold Rise of anti-OspA Binding IgG Antibody Concentration at Days 29, 85, and 197 Compared to Day 1 (Baseline) | Days 29, 85, and 197

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Encore Research Group-Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Clinical Research-DeLand, LLC d/b/a Accel Research Sites, Lake Mary, Florida
  - Clinical Research Atlanta, headlands LLC, Stockbridge, Georgia
  - Johnson County Clin-Trials, Inc. (JCCT), Lenexa, Kansas
  - Centennial Medical Group, Columbia, Maryland
  - Advanced Primary and Geriatric Care, Rockville, Maryland
  - DM Clinical Research - Brookline, Brookline, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Meridian Clinical Research - Omaha, Omaha, Nebraska
  - ActivMed Research LLC, Newington, New Hampshire
  - Rochester Clinical Research, Inc., Rochester, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Hatboro Medical Associates/CCT Research, Hatboro, Pennsylvania
  - Velocity Clinical Research Providence, Providence, Rhode Island
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research, Tomball, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia